CLINICAL TRIAL: NCT06774261
Title: A Phase 1b Dose Range Finding Study of Phenserine Compared to Donepezil in Participants With Early or Mild Alzheimer's Disease
Brief Title: Phenserine on the Alzheimer's Treatment Horizon, Study 1
Acronym: PATH-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Fonna (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); University of Exeter (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EuCT: 2023-510282-10-00
Record Dates: First submitted 2024-10-18; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Alzheimer's Disease; Phenserine; Donepezil; Randomized Controlled Trial; Cognitive Decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — phenserine; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenserine (Active Comparator): Phenserine will be formulated as a capsule, with dosages of 5mg and 10mg. Participants randomized to the phenserine arm will start at 5 mg twice daily (bd) with escalations every two weeks, as tolerated to 10 mg bd and to a maximum dose of 10 mg three times daily (tds).
  Interventions: Drug: Phenserine
- Donepezil (Active Comparator): Participants randomized to the donepezil arm will start at 5 mg tablet once daily (od) with escalation, to 10 mg od from Week 5, as tolerated.
  Interventions: Drug: Donepezil (Aricept®)

INTERVENTIONS:
Drug: Phenserine — Phenserine is a next generation AChE inhibitor being developed for the treatment of AD. Unlike currently marketed AChE inhibitors, it has additional mechanisms of action that also include a mediating effect on cell death pathways and anti-amyloid activity, which may confer disease-modifying effects in people with AD.
  Phenserine was originally identified and developed by the United States (U.S.) National Institute of Aging (NIA), part of the U.S National Institute of Health (NIH).
  The study intervention will be open label. No blinding will be performed. Participants and site staff will, however, will be blinded to the results of the exosome and blood/CSF biomarker evaluations until the study is completed.
  Arms: Phenserine
Drug: Donepezil (Aricept®) — The substance donepezil (under the brand name Aricept®) is a resale product. No additional manufacturing or labeling measures is necessary for this study.
  The NIMP, donepezil will be available in 5 mg and 10 mg strengths (table 3) and will be dispensed by the local pharmacy at the hospital where the participant in the donepezil arm is included. We have based the use of donepezil as a treatment in the study on the original product from Pfizer, but it is also possible to use generic products of donepezil if this is what the local pharmacy has for dispensing. Participants randomized to treatment with donepezil will follow the treatment plan according to the patient information leaflet. . These tablets are approved for clinical use and comply with all relevant safety and efficacy standards.
  Arms: Donepezil

SUMMARY:
The goal of this clinical trial is to evaluate if phenserine can treat early or mild Alzheimer's Disease (AD) by comparing it to donepezil. This study will include participants with early or mild Alzheimer's Disease, and the main questions it aims to answer are:

How does phenserine affect exosome biomarkers of cell death compared to donepezil? What is the safety and tolerability profile of phenserine at ascending oral doses compared to donepezil? Researchers will compare participants receiving phenserine to those receiving donepezil to see if phenserine produces better pharmacodynamic outcomes and if it is safe and well-tolerated.

Participants will:

Be randomized to receive either oral phenserine or oral donepezil for a treatment duration of 8 weeks.

Undergo oral dose escalation based on tolerability. Complete regular follow-up visits every two weeks to assess pharmacodynamic, pharmacokinetic, and safety measures.

DETAILED DESCRIPTION:
Participants will be randomized into two groups: one group will receive phenserine, and the other will receive donepezil. The phenserine group will begin with a dosage of 5 mg twice daily, with the dose being gradually increased every two weeks as tolerated with a maximum dose of 10 mg three times daily. The donepezil group will start at 5 mg once daily, with the possibility of escalation to 10 mg once daily at Week 4.

The study is designed to last 8 weeks, with a planned total enrollment of 16 individuals from various centers across Norway. Participants will return for follow-up visits every two weeks, during which pharmacodynamic, pharmacokinetic, and safety assessments will be conducted. The final safety follow-up will occur after the completion of dosing for those who complete the study. Early termination visits will include a comprehensive safety follow-up for those who discontinue the study prematurely.

The primary objective of this study is to assess the effects of phenserine compared to donepezil on exosome biomarkers of cell death in individuals with early or mild AD. Additionally, the study aims to evaluate the safety and tolerability profile of phenserine at ascending doses up to 10 mg three times daily (QDS) in comparison to donepezil at doses up to 10 mg once daily (OD). Furthermore, the study aims to analyze steady-state blood levels of phenserine to characterize and compare dose-response relationships for pharmacodynamic outcomes and key safety assessments. Finally, the study will explore changes in specific biomarkers of Alzheimer's Disease (AD) in cerebrospinal fluid (CSF) and blood plasma, as well as assess phenserine's potential short-term effects on cognition using the FLAME Memory Composite and other cognitive sub-tests.

Participants will be enrolled at six centers across Norway. The study will also be supported by the PROTECT platform, which allows for the recruitment of individuals over 50 years of age who have demonstrated cognitive decline, making them suitable candidates for this study.

The anticipated duration of participation for each patient is 8 weeks, with the overall study expected to be completed within 9 months, accounting for a 6-month enrollment period followed by the treatment phase.

Study Population and Statistical Methods

A total of 16 participants are expected to be enrolled in this dose-ranging study. The primary population for analysis will be a modified intent-to-treat group, including all participants who received at least one dose of study medication and provided at least one follow-up exosome sample.

This study will provide critical data on the pharmacodynamic and pharmacokinetic profiles of phenserine, which will guide future research and potential therapeutic strategies for early to mild AD.

Background

In 2018, and in parallel with the conduct of the ELAD study that evaluated liraglutide (an established medication for Type 2 diabetes) for its neuroprotective effects in people with mild to moderate AD, we initiated a new selection process to identify additional drug candidates for re-purposing in AD, MCI and other forms of dementia. Drug repurposing, defined as "the application of established drug compounds to new therapeutic indications," offers a route to drug development that is accessible to academic institutions, government and research council programs, and charities and not-for-profit organizations, complementing the work of pharmaceutical and biotechnology companies. Repurposing an existing drug offers an attractive way of enhancing traditional drug development and accelerating new treatments for people with AD dementia and MCI into the clinic.

The international expert panel that participated in the 2018 assessment applied the same approach as in the earlier 2012 selection process. A total of five compounds or classes of compounds were nominated for further consideration by the panel. These compounds were ACE inhibitors, antiviral drugs, disease-modifying antirheumatic drugs (DMARDs), fasudil and phenserine. Following several rounds of prioritization, the panel came to a clear consensus that the three highest priority candidates for repurposing in AD, MCI and other dementias were phenserine, fasudil, and antiviral drugs. This protocol is designed to assess the safety and tolerability of phenserine compared to donepezil across a range of doses administered over a 8-week dosing period in participants with early or mild AD. The pharmacodynamic and pharmacokinetic activity of the two drugs will also be evaluated to determine dose-response relationships to identify an appropriate dose range for a subsequent Phase 2 study of phenserine.

Phenserine was initially developed as an acetylcholinesterase inhibitor (AChEI) , but there are several mechanisms by which phenserine may act on neuronal and synaptic loss , a key common pathway evident in AD. A range of pre-clinical studies indicate that phenserine suppresses interleukin-1b, reduces glutamate-induced excitotoxicity, protects against oxidative toxicity, reduces A-beta levels, improves neural precursor cell viability, elevates neurotrophic brain-derived neurotrophic factor, and inhibits amyloid-beta precursor protein synthesis. In the only published phase 2 randomized controlled trial (RCT), phenserine (10-15 mg b.i.d.) conferred improvement in cognition in people with AD receiving 12 weeks of the higher dose of phenserine. Safety and tolerability were very good. The proportion of withdrawals due to adverse events was 6% in the placebo arm and the highest dose groups, indicating that the optimal dose was probably not achieved for most patients. There were also methodological problems, prompting the authors to conclude that the full potential of phenserine for AD has not yet been fully evaluated.

The most common side-effects of phenserine are those associated with cholinesterase inhibition, i.e., nausea, vomiting and diarrhoea. The best predictor of cholinesterase linked gastrointestinal effects is the level of cholinesterase inhibition achieved, with the optimal therapeutic threshold being 50% inhibition. Given that the completed clinical trials with phenserine did not select patients based on biomarker confirmation of AD (meaning that a considerable proportion of participants likely did not have AD), and that the maximum dose did not lead to side-effects and thus many participants did not likely achieve a sufficiently high dose level, this study aims to evaluate the effects of an individualized maximum tolerated phenserine dose with adequate level of AChE inhibition to determine an appropriate dose range for subsequent efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of AD based on the most recent NIA-AA diagnostic criteria for AD.
* A significant change on a validated AD amyloid or tau biomarker (as determined either by visual reading of amyloid PET scans [using any of the approved ligands], or CSF Aβ 1-42 or blood p-tau 217 levels [cut-off as determined by the individual laboratory.
* A CDR Global rating of 0.5 or 1.0.
* An MRI scan within the past two years that has no findings inconsistent with AD.
* Participants who have recently participated in other clinical trials or have been under treatment with memantine or acetylcholinesterase inhibitors (e.g., Donepezil, Rivastigmine, Galantamine) must undergo a washout period of at least 4 weeks prior to the start of the study.
* Capacity to give informed consent based on the clinical judgement of an experienced clinician.
* The participant has an individual who is in regular, daily contact via phone or in-person visits and who can act as a reliable study partner and provide meaningful input into rating scales.
* Age ≥50 years.
* Fluency in Norwegian and evidence of adequate premorbid intellectual functioning.
* Capable of participating in all scheduled evaluations and complete all required tests.
* Female participants must be of non-childbearing potential or have a negative serum pregnancy test up to 24 hours prior to the baseline assessments and agree to use effective birth control throughout their participation in the study from signing informed consent form until at least 30 days after last administration of phenserine or donepezil..

Exclusion Criteria:

* Significant cerebrovascular disease, as indicated by clinical history, neurological examination, or on MRI (including cortical infarction or deep white matter or periventricular white matter hyperintensities with a Fazekas scale score of 3 (25).
* Current treatment with a cholinesterase inhibitor or memantine.
* Hypersensitivity to AChE inhibitors or related compounds: Known hypersensitivity to donepezil, piperidine derivatives, or any formulation components.
* Participants undergoing or planning procedures requiring anesthesia with depolarizing neuromuscular blockers (e.g., succinylcholine) due to the risk of prolonged paralysis or apnea when combined with AChE inhibitors.
* Active peptic ulcer disease or gastrointestinal bleeding, or a history of gastrointestinal ulcers or bleeding.
* Severe cardiac conditions: Significant arrhythmias, sick sinus syndrome, supraventricular conduction abnormalities, or other cardiac rhythm disorders that could pose a risk with cholinesterase inhibitors.
* Severe respiratory disease: Chronic obstructive pulmonary disease (COPD) or poorly controlled asthma.
* History of urinary obstruction or bladder issues, particularly those requiring catheterization.
* Current clinically significant depression or other mental disorders likely to affect cognition or interfere with study participation.
* Participants using sedating drugs, if unavoidable, will be excluded from the study. However, short-acting sleep medications can be used if taken as recommended and if the participant has maintained a stable regimen for at least 3 months prior to the start of the study.
* Current participation in any other drug trial(s).
* Currently ongoing life-threatening disease, such as metastatic cancer, advanced cardiovascular disease, advanced respiratory disease, terminal kidney disease, or advanced stages of an infectious disease.
* Any current or past neurological disease unrelated to AD and with cognitive sequelae.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Panel 1: Concentration of Biomarkers Associated with Preprogrammed Cell Death (PNCDD) | From enrollment to the end of treatment at 8 weeks.
  Quantification of exosome-derived BAX and Bcl-2 markers. This outcome measure will assess changes in biomarkers related to preprogrammed cell death, specifically BAX and Bcl-2. These biomarkers provide insights into apoptotic processes and any alterations observed following treatment with phenserine or donepezil.
Panel 2: Concentration of Synaptic Integrity Biomarkers | From enrollment to the end of treatment at 8 weeks.
  Measurement of exosome-derived synaptic markers. This outcome measure will evaluate changes in synaptic markers, including synaptotagmin, to provide insights into synaptic integrity and function.
Panel 3: Concentration of TNF-α (Inflammatory Biomarker) | From enrollment to the end of treatment at 8 weeks.
  Quantification of exosome-derived TNF-α. This outcome measure will assess changes in TNF-α levels (ng/mL), a key inflammatory biomarker.
Panel 3: Concentration of interleukins, IL-1β, IL-6, and IL-10. (Inflammatory Biomarker) | From enrollment to the end of treatment at 8 weeks.
  Quantification of exosome-derived IL-1β, IL-6, and IL-10.IL-1β (pg/mL). This outcome measure will assess changes in interleukin levels, a key inflammatory biomarker.
Panel 4: Concentration of Exosome-Derived Alzheimer's Disease-Specific Biomarkers | From enrollment to the end of treatment at 8 weeks.
  Quantification of exosome-derived Aβ1-42. This outcome measure will assess changes in exosome-derived Alzheimer's Disease-specific biomarkers, including Aβ1-42, to elucidate molecular signatures associated with AD pathology.

SECONDARY OUTCOMES:
Adverse Events (AEs) and Tolerability Profile | From enrollment to the end of treatment at 8 weeks.
  Safety and tolerability will be evaluated based on reported or observed adverse events (AEs), including those related to acetylcholinesterase inhibitors (AChEI). The frequency, severity, and relationship of AEs to treatment will be documented throughout the study. The unit of measure will be the number of participants experiencing AEs.
Cholinesterase Inhibition Target Achievement | From enrollment to the end of treatment at 8 weeks.
  Percentage of participants achieving target inhibition (%), time to target (days), and duration of inhibition (days).The proportion of participants in the phenserine arm achieving the target cholinesterase inhibition of ~45% will be evaluated, along with the time to reach this target and duration of maintaining the inhibition.
Blood Pressure (Safety Assessment) | From enrollment to the end of treatment at 8 weeks
  Blood pressure measured in millimeters of mercury (mmHg).
Pulse (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Pulse (Safety Assessment). Pulse frequency measured in beats per minute (bpm).
Urine Testing (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Urine will be tested with a dipstick to explore proteinuria or hematuria.
Blood Urea Nitrogen (BUN) (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Blood Urea Nitrogen (BUN) (Safety Assessment). Measured in blood in mmol/L.
Potassium (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in mmol/L.
Sodium (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in mmol/L.
Calcium (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in mmol/L.
Glucose (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in mmol/L.
Creatinine (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in μmol/L.
Total and Direct Bilirubin (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in μmol/.
C-Reactive Protein (CRP) (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measured in blood in mg/L.
Liver function (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase. Measured in blood in U/L.
Electrocardiogram (ECG) (Safety Assessment) | From enrollment to the end of treatment at 8 weeks.
  Measurement of ECG QT Interval. Measured in ms (milliseconds).
Columbia Suicide Severity Rating Scale (C-SSRS) (Safety Assessment) | At enrollment, week 4 and of treatment at 8 weeks.
  Participants will be monitored for suicidal ideation and unusual behavior using the C-SSRS.
Maximum Plasma Concentration (Cmax) of Phenserine | Measured at week 2, week 4, week 6 and of treatment at 8 weeks.
  Plasma samples will be analyzed to determine the maximum plasma concentration (Cmax) of phenserine.
Half-Life (t1/2) of Phenserine and Donepezil | Measured at week 2, week 4, week 6 and of treatment at 8 weeks.
  Plasma samples will be used to determine the half-life (t1/2) of phenserine and donepezil, representing the time it takes for the drug's plasma concentration to reduce by half.
Steady-State Concentration of Phenserine and Donepezil | Measured at week 2, week 4, week 6 and of treatment at 8 weeks.
  Plasma samples collected at Week 8 (at peak dose) from all participants, or at the final maintenance dose for those who down-titrate, will be used to evaluate the steady-state concentration of phenserine and donepezil.

OTHER OUTCOMES:
FLAME computer-based domain composites | At baseline and end of treatment at 8 weeks
  Neuropsychology assessments will be conducted using the FLAME computer-based domain composites for memory, executive function, attention and sustained attention to evaluate changes over the 10-week treatment period in the phenserine-treated participants compared to those who received donepezil. The results of these assessments will be compared to changes observed on exosome biomarkers to identify similar trends across the treatment arms and in individual participants.
Montreal Cognitive Assessment (MoCA) | At baseline and end of treatment at 8 weeks.
  The Montreal Cognitive Assessment (MoCA) will be used at baseline and end-of-treatment to assess for any changes in cognition over the course of the treatment period. The MoCA score ranges from 0 to 30, with higher scores indicating better cognitive performance.
Cerebrospinal Fluid (CSF) Levels of Aβ1-40 and Aβ1-42 | Baseline and end of treatment at 8 weeks.
  CSF samples will be collected and analyzed for amyloid-beta (Aβ1-40 and Aβ1-42), key biomarkers of Alzheimer's Disease (AD) pathology. Units of Measure: pg/mL.
Cerebrospinal Fluid (CSF) Levels of Total Tau (tTau) and Phosphorylated Tau (pTau) | Baseline and end of treatment at 8 weeks.
  CSF samples will be collected and analyzed for total tau (tTau) and phosphorylated tau (pTau), markers of neurofibrillary tangles and AD-specific pathology. Units of Measure: pg/mL.
Plasma Levels of pTau217 | Baseline and end of treatment at 8 weeks.
  Plasma samples will be collected and analyzed for levels of phosphorylated tau (pTau217), a biomarker associated with Alzheimer's Disease (AD) pathology. Units of Measure: pg/mL.
Plasma Levels of Neurofilament Light Chain (NfL) | Baseline and end of treatment at 8 weeks.
  Plasma samples will be collected and analyzed for levels of neurofilament light chain (NfL), a biomarker of neurodegeneration in Alzheimer's Disease (AD). Units of Measure: pg/mL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reijs BL, Teunissen CE, Goncharenko N, Betsou F, Blennow K, Baldeiras I, Brosseron F, Cavedo E, Fladby T, Froelich L, Gabryelewicz T, Gurvit H, Kapaki E, Koson P, Kulic L, Lehmann S, Lewczuk P, Lleo A, Maetzler W, de Mendonca A, Miller AM, Molinuevo JL, Mollenhauer B, Parnetti L, Rot U, Schneider A, Simonsen AH, Tagliavini F, Tsolaki M, Verbeek MM, Verhey FR, Zboch M, Winblad B, Scheltens P, Zetterberg H, Visser PJ. The Central Biobank and Virtual Biobank of BIOMARKAPD: A Resource for Studies on Neurodegenerative Diseases. Front Neurol. 2015 Oct 15;6:216. doi: 10.3389/fneur.2015.00216. eCollection 2015. PMID 26528237
- [Background] Tweedie D, Fukui K, Li Y, Yu QS, Barak S, Tamargo IA, Rubovitch V, Holloway HW, Lehrmann E, Wood WH 3rd, Zhang Y, Becker KG, Perez E, Van Praag H, Luo Y, Hoffer BJ, Becker RE, Pick CG, Greig NH. Cognitive Impairments Induced by Concussive Mild Traumatic Brain Injury in Mouse Are Ameliorated by Treatment with Phenserine via Multiple Non-Cholinergic and Cholinergic Mechanisms. PLoS One. 2016 Jun 2;11(6):e0156493. doi: 10.1371/journal.pone.0156493. eCollection 2016. PMID 27254111
- [Background] Greig NH, De Micheli E, Holloway HW, Yu QS, Utsuki T, Perry TA, Brossi A, Ingram DK, Deutsch J, Lahiri DK, Soncrant TT. The experimental Alzheimer drug phenserine: preclinical pharmacokinetics and pharmacodynamics. Acta Neurol Scand Suppl. 2000;176:74-84. doi: 10.1034/j.1600-0404.2000.00311.x. PMID 11261809
- [Background] Chang CF, Lai JH, Wu JC, Greig NH, Becker RE, Luo Y, Chen YH, Kang SJ, Chiang YH, Chen KY. (-)-Phenserine inhibits neuronal apoptosis following ischemia/reperfusion injury. Brain Res. 2017 Dec 15;1677:118-128. doi: 10.1016/j.brainres.2017.09.015. Epub 2017 Sep 27. PMID 28963051
- [Background] Becker RE, Greig NH, Giacobini E, Schneider LS, Ferrucci L. A new roadmap for drug development for Alzheimer's disease. Nat Rev Drug Discov. 2014 Feb;13(2):156. doi: 10.1038/nrd3842-c2. Epub 2013 Dec 20. No abstract available. PMID 24362362
- [Background] Braida D, Sala M. Eptastigmine: ten years of pharmacology, toxicology, pharmacokinetic, and clinical studies. CNS Drug Rev. 2001 Winter;7(4):369-86. doi: 10.1111/j.1527-3458.2001.tb00205.x. PMID 11830755
- [Background] Desai A, Grossberg G. Review of rivastigmine and its clinical applications in Alzheimer's disease and related disorders. Expert Opin Pharmacother. 2001 Apr;2(4):653-66. doi: 10.1517/14656566.2.4.653. PMID 11336614
- [Background] Wilkinson DG, Francis PT, Schwam E, Payne-Parrish J. Cholinesterase inhibitors used in the treatment of Alzheimer's disease: the relationship between pharmacological effects and clinical efficacy. Drugs Aging. 2004;21(7):453-78. doi: 10.2165/00002512-200421070-00004. PMID 15132713
- [Background] Nordberg A, Kadir A, Andreasen N, Almkvist O, Wall A, Langstrom B, Zetterberg H. Correlations between Alzheimer's Disease Cerebrospinal Fluid Biomarkers and Cerebral Glucose Metabolism after 12 Months of Phenserine Treatment. J Alzheimers Dis. 2015;47(3):691-704. doi: 10.3233/JAD-132474. PMID 26401704
- [Background] Kadir A, Andreasen N, Almkvist O, Wall A, Forsberg A, Engler H, Hagman G, Larksater M, Winblad B, Zetterberg H, Blennow K, Langstrom B, Nordberg A. Effect of phenserine treatment on brain functional activity and amyloid in Alzheimer's disease. Ann Neurol. 2008 May;63(5):621-31. doi: 10.1002/ana.21345. PMID 18300284
- [Background] Becker RE, Greig NH, Lahiri DK, Bledsoe J, Majercik S, Ballard C, Aarsland D, Schneider LS, Flanagan D, Govindarajan R, Sano M, Ferrucci L, Kapogiannis D. (-)-Phenserine and Inhibiting Pre-Programmed Cell Death: In Pursuit of a Novel Intervention for Alzheimer's Disease. Curr Alzheimer Res. 2018;15(9):883-891. doi: 10.2174/1567205015666180110120026. PMID 29318971
- [Background] Greig NH, Ruckle J, Comer P, Brownell L, Holloway HW, Flanagan DR Jr, Canfield CJ, Burford RG. Anticholinesterase and pharmacokinetic profile of phenserine in healthy elderly human subjects. Curr Alzheimer Res. 2005 Oct;2(4):483-92. doi: 10.2174/156720505774330564. PMID 16248851